CLINICAL TRIAL: NCT00374699
Title: A Phase I/II Study of Bortezomib + CHOP in Patients With Advanced Stage Aggressive T Cell or NK/T Cell Lymphomas
Brief Title: Bortezomib and CHOP in Patients With Advanced Stage Aggressive T Cell or Natural Killer (NK)/T Cell Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Janssen Medical Affairs (Industry)
Responsible Party: CISL (Consortium for Improving Survival of Lymphoma), CISL (Consortium for Improving Survival of Lymphoma)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-07-021
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2007-06

CONDITIONS: Peripheral T-Cell Lymphomas; Non-Hodgkin Lymphoma
Keywords: Velcade; Bortezomib; CHOP; Peripheral T-cell lymphomas(PTCLs); natural killer (NK)-cell lymphomas
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Non-Hodgkin | interventions — Bortezomib

INTERVENTIONS:
Drug: Velcade

SUMMARY:
Peripheral T-cell lymphomas (PTCLs) are neoplasias from post-thymic T-cells at different stages of differentiation and are a heterogeneous group of malignancies which present with different morphological patterns, phenotypes, and clinical presentations.

These tumours have a striking epidemiological distribution with a lower incidence in Western countries than in Asia. In Korea, PTCLs including T- or natural killer (NK)-cell lymphomas constitute approximately 25 to 35% of all non-Hodgkin's lymphomas. This incidence is quite similar to that of other Eastern Asian countries, including Japan, Hong Kong, and China.

Recent studies suggest that the T-cell phenotype is an independent significant prognostic factor, with PTCLs having one of the lowest overall survival and failure-free survival rates. Based on the investigator's experience, the overall complete remission rate was 61.2% (95% confidence interval [CI]: 48.5-72.8%) and the 5-year probability of failure-free survival was 33.5%. Median survival of all patients was 45 months (range 0-64+ months) and the 5-year probability of survival was 36.2%. Rassidakis et al. reported that expression of pro-apoptotic proteins BAX and BCL-XS, may explain the poor response of many types of PTCL to standard chemotherapy.

To overcome such poor outcome, the optimal therapy for PTCLs remains to be defined. However, because of the rarity of the disease in Western countries, only a few trials have been reported.

Bortezomib (Velcade) is a modified dipeptidyl boronic acid, and a reversible inhibitor of the chymotrypsin-like activity of the 26S proteosome. Bortezomib may induce tumor cell apoptosis or decreased bcl-2 associated drug resistance. Through phase II studies, single agent bortezomib in patients with relapsed indolent and mantle cell lymphomas showed its activity. And also preliminary data indicate that bortezomib can be safely administered in combination with dose adjusted etoposide, prednisolone, vincristine, cyclophosphamide and doxorubicin (EPOCH) chemotherapy. Therefore, it can be possible to improve the poor outcome of patients with PTCLs by a combination of cyclophosphamide, doxorubicin, vincristine, prednisolone (CHOP) with bortezomib as a first-line therapy.

Primary Hypothesis: Based on the clinical trials and experimental data, bortezomib can overcome pro-apoptotic proteins BAX and BCL-XS induced drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed PTCLs and NK/T cell lymphomas excluding anaplastic lymphoma kinase (ALK)-positive anaplastic large cell T-cell lymphomas (ALCL)
* Performance status (ECOG) ≤ 3
* Age ≤ 65
* At least one or more unidimensionally measurable lesion(s)

  * ≥ 2 cm by conventional computed tomography (CT)
  * ≥ 1 cm by spiral CT
  * skin lesion (photographs should be taken)
  * measurable lesion by physical examination
* Laboratory values

  * Creatinine (Cr) < 1.5 mg% or creatinine clearance (Ccr) > 50 ml/min
  * Transaminase < 3 X upper normal value
  * Bilirubin < 2.0 mg/dl
  * Absolute neutrophil count (ANC) > 1,500/ul
  * Platelets > 75,000/ul
* Informed consent
* Ann Arbor stage III or IV

Exclusion Criteria:

* Any other malignancies within the past 5 years except basal cell skin cancer or carcinoma in situ (CIS) of the cervix
* Serious comorbid diseases
* Pregnancy or breast feeding

Any waiver of these inclusion and exclusion criteria must be approved by the investigator and the sponsor on a case-by-case basis prior to enrolling the subject. This must be documented by both the sponsor and the investigator. No subject will be allowed to enroll in this study more than once.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To define the dose-limiting toxicity and maximum tolerable dose | Phase I
To evaluate the overall response rate | Phase II

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the treatment combination | Phase I/II
To estimate the time to progression and the duration of overall response | Phase II

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea